CLINICAL TRIAL: NCT06947551
Title: The Mechanism of Endogenous Nociceptin/Orphanin FQ(N/OFQ) and β1-adrenoceptor Autoantibody in Promoting Ischemic Arrhythmia in Rats
Acronym: tmoenabaaipiai
Status: Not yet recruiting | Type: Observational
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, Professor, Second Hospital of Shanxi Medical University
Other Study IDs: HY20240410
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with coronary heart disease or diabetes under different course of disease: Select patients with coronary heart disease and diabetes who meet the standard, take 8ml of blood from the elbow vein, 4ml of blood for centrifugation, take serum, and use chromatography column to separate and extract β 1-AA; 4ml is used to detect endogenous N/OFQ and β 1-AA levels using an ELISA kit.

SUMMARY:
In the early stage of ischemic arrhythmia, endogenous N/OFQ regulates the expression of β 1-AA, mediates the internalization of β 1-AR by PKC/ERK1/2, and thus affects the occurrence of arrhythmia. Further clarify the regulatory mechanism of N/OFQ on β 1-AR internalization and arrhythmia, providing experimental basis for drug development and target exploration of clinical ischemic arrhythmia; To observe the relationship between endogenous N/OFQ and β 1-AA in serum of patients with coronary heart disease and diabetes.

DETAILED DESCRIPTION:
This project mainly involves animal experiments and cell experiments. The part of clinical trials involved is the extraction of autoantibodies to β 1-adrenoceptor (β 1-AA) from the serum of patients with coronary heart disease and diabetes. The purified antibodies are intended to be used as agonists to rapidly increase the concentration of β 1-AA in the body of animals and the environment of cells in a short time, observe the impact of the antibodies on animals and cells, and further clarify that β 1-AA affects the internalization of β 1-AR through PKC/ERK1/2 at the early stage of blood arrhythmia, so as to regulate the occurrence of arrhythmia. After reviewing the literature, we found that β 1-AA exists in patients with ischemic arrhythmia, coronary heart disease, dilated cardiomyopathy, heart failure, diabetes, dogs with dilated heart disease and hypertensive rats. These β 1-AA targets the second extracellular ring of β 1-AR. Moreover, it can produce an agonist like response to spontaneously beating rat cardiomyocytes, inducing ventricular arrhythmias by stimulating β 1-AR and its downstream pathways. This experiment plans to select 60 patients and extract 8ml and 4ml of blood from the elbow vein for centrifugation and serum extraction. β 1-AA will be separated and extracted using a chromatography column; 4ml is used to detect endogenous N/OFQ and β 1-AA levels using an ELISA kit.

ELIGIBILITY:
Inclusion Criteria:1) Inclusion criteria for patients with diabetes: refer to the diagnostic criteria for type 2 diabetes (T2DM) in the Chinese Guidelines for the Prevention and Treatment of Type 2 diabetes (2017) 2) Inclusion criteria for patients with coronary heart disease: patients with clinically diagnosed coronary heart disease according to the 1979 WHO Diagnostic Criteria for Ischemic Heart Disease, and exclusion criteria include heart failure, tumor, immune disease and diabetes. -

Exclusion Criteria:Exclusion criteria for patients with coronary heart disease: including heart failure, tumor, immune disease and diabetes. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart disease or diabetes under different course of disease
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Orphanin and β 1-AA in Serum of Patients with Coronary Heart Disease or diabetes of Different Course | The patient's first blood draw upon admission
  To measure the content of orphanin and β 1-AA in the serum of patients with coronary heart disease or diabetes of different disease courses, and to explore the relationship between orphanin and β 1-AA in the serum of patients with different disease courses, so as to provide support for the prediction of clinical coronary heart disease or diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: yi Han, Study Director — Second Hospital of Shanxi Medical University

IPD SHARING:
Plan to Share IPD: No